CLINICAL TRIAL: NCT01172132
Title: Long Term Outcomes in Critically Ill Haematological Patients. The Use of Intensive Care in Critically Ill Cancer Haematological Patients
Brief Title: The Use of Intensive Care in Critically Ill Cancer Haematological Patients: "TRIAL-OH"
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM 08235
Record Dates: First submitted 2010-06-18; First posted 2010-07-29 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2011-11

CONDITIONS: Hematological Malignancies
Keywords: Leukemia; Lymphoma; Bone-Marrow Transplant; Neutropenia; Acute respiratory failure; Mechanical ventilation; Post ICU burden; ICU triage; Dialysis; Septic shock
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Neutropenia; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine:

* Condition of intensive care unit (ICU) admission in patients with haematological malignancies.
* ICU hospital and up to one year mortality.
* Assessment of post ICU burden and health related quality at 90-d and 1 year.

DETAILED DESCRIPTION:
1. To identify prognostic factors of short and medium term mortality, by underlining the respective weights of organ dysfunction and characteristics of underlined malignancy
2. Evaluate the health related quality of life of intensive care survivors(SF36)
3. Impact of intensive care on families burden (HADS, IES).
4. Assess clinicians' satisfaction ( intensivists, haematologists and intensive care nurses) in relation to medical decision-making.
5. Establish the relevance of antifungal treatments.

ELIGIBILITY:
Inclusion Criteria:

* Hematological malignancies
* hospitalization in ICU
* age >= 18 years

Exclusion Criteria:

* Patients who have already participated to TRIAL-OH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heamatological malignancy adressed to ICU
Sampling Method: Probability Sample
Enrollment: 1011 (Actual)
Dates: Start 2009-11; Primary Completion 2011-05 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Survival status at one year | 1 year
  survival status (alive or death) at one year

SECONDARY OUTCOMES:
Health related quality of life of patients and their relatives | day 90 and 1 year
ICU mortality | 1 week (estimated mean time until ICU discharge)
  survival status at ICU discharge
Survival status | day 90
Hospital mortality | 3 weeks (estimated mean time until Hospital discharge)
  survival status at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Elie Azoulay, MD, PhD, Principal Investigator — Saint-Louis Hospital, Paris, France
Locations (1):
- Hôpital Saint-Louis, AP-HP, Paris, France

REFERENCES:
- [Background] Camous L, Lemiale V, Canet E, Max A, Schnell D, Le Goff J, Rabbat A, Schlemmer B, Azoulay E. Clinical features of H1N1 2009 infection in critically ill immunocompromised patients. Crit Care. 2010;14(2):139. doi: 10.1186/cc8927. Epub 2010 Apr 14. PMID 20392286
- [Result] Lemiale V, Resche-Rigon M, Mokart D, Pene F, Rabbat A, Kouatchet A, Vincent F, Bruneel F, Nyunga M, Lebert C, Perez P, Meert AP, Benoit D, Chevret S, Azoulay E. Acute respiratory failure in patients with hematological malignancies: outcomes according to initial ventilation strategy. A groupe de recherche respiratoire en reanimation onco-hematologique (Grrr-OH) study. Ann Intensive Care. 2015 Dec;5(1):28. doi: 10.1186/s13613-015-0070-z. Epub 2015 Sep 30. PMID 26429355
- [Derived] Zafrani L, Resche-Rigon M, De Freitas Caires N, Gaudet A, Mathieu D, Parmentier-Decrucq E, Lemiale V, Mokart D, Pene F, Kouatchet A, Mayaux J, Vincent F, N'yunga M, Bruneel F, Rabbat A, Lebert C, Perez P, Meert AP, Benoit D, Darmon M, Azoulay E. Endothelial Cell-Specific Molecule-1 in Critically Ill Patients With Hematologic Malignancy. Crit Care Med. 2018 Mar;46(3):e250-e257. doi: 10.1097/CCM.0000000000002934. PMID 29474336
- [Derived] Contejean A, Lemiale V, Resche-Rigon M, Mokart D, Pene F, Kouatchet A, Mayaux J, Vincent F, Nyunga M, Bruneel F, Rabbat A, Perez P, Meert AP, Benoit D, Hamidfar R, Darmon M, Jourdain M, Renault A, Schlemmer B, Azoulay E. Increased mortality in hematological malignancy patients with acute respiratory failure from undetermined etiology: a Groupe de Recherche en Reanimation Respiratoire en Onco-Hematologique (Grrr-OH) study. Ann Intensive Care. 2016 Dec;6(1):102. doi: 10.1186/s13613-016-0202-0. Epub 2016 Oct 25. PMID 27783381